CLINICAL TRIAL: NCT00937846
Title: An Open Label Positron Emission Tomography (PET) Study to Investigate Brain Penetration by [Carbonyl-11C] GSK1034702 in Healthy Subjects
Brief Title: Brain Uptake of GSK1034702: a Positron Emission Tomography (PET) Scan Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 110771
Record Dates: First submitted 2009-06-25; First posted 2009-07-13 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Cognitive Disorders
Keywords: Cognitive impairment; Schizophrenia; Alzheimer's Disease; PET
MeSH Terms: conditions — Cognitive Dysfunction; Schizophrenia; Alzheimer Disease | interventions — GSK 1034702

ARMS (1):
- GSK1034702 (Experimental): Single oral 5 mg dose in liquid formulation
  Interventions: Drug: GSK1034702

INTERVENTIONS:
Drug: GSK1034702 — Single oral 5 mg dose in liquid formulation

SUMMARY:
GSK1034702 is being developed for improving cognitive impairment in diseases such as Alzheimer's disease and schizophrenia. This study will be done in healthy men to investigate how much of the study drug gets into the brain. This will be done using Positron Emission Tomography (PET).

DETAILED DESCRIPTION:
This is an open label, single dose, non-randomized PET study in healthy male subjects to ascertain if GSK1034702 is crossing the blood-brain barrier to enable it to elicit a central effect. GSK1034702 has been shown in vitro to be a substrate for human Pgp, therefore the distribution of GSK1034702 into human brain could be adversely affected. This use of PET in conjunction with radioactively labelled GSK1034702 will help ascertain the role Pgp plays in limiting brain penetration in the presence and absence of a pharmacological relevant oral non labelled dose of 5 mg. Subjects will have an MRI scan to aid definition of brain anatomy, a baseline PET scan and a post-dose PET scan. For each subject the study will consist of at least three visits; screening visit, scanning day and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy.
* Male between 35 and 55 years of age.
* Willing to use appropriate contraception method.
* Weight more than 50 kg.
* BMI within the range 19 - 29 kg/m2.
* Adequate blood supply to the hand.

Exclusion Criteria:

* Abuse of drugs or alcohol.
* Smoker or history of regular use of tobacco- or nicotine-containing products in the past 6 months.
* ECG abnormality (personal or family history).
* Psychiatric disorder.
* Asthma or a history of asthma.
* Medical illness.
* Worked as a welder, metal worker or machinist.
* Suffers from claustrophobia or would be unable to lie still in a PET or MRI scanner for 1-2 hours.
* Has a cardiac pacemaker or other electrical device or ferromagnetic metal foreign bodies.
* Neurological disorder

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2009-07-15 (Actual); Primary Completion 2009-08-28 (Actual); Study Completion 2009-08-28 (Actual)

PRIMARY OUTCOMES:
Volume of distribution of [11C]GSK1034702 at tracer and pharmacological doses. | Scanning day

SECONDARY OUTCOMES:
The kinetic rate constants at tracer and pharmacological doses. | Scanning day
GSK1034702 PK parameters: Cmax; tmax; AUC(0-t). | Scanning day
Safety and tolerability endpoints consisting of: AEs; 12-lead ECG; 12 lead digital Holter and lead II telemetry; vital signs; clinical laboratory evaluations. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Ridler K, Cunningham V, Huiban M, Martarello L, Pampols-Maso S, Passchier J, Gunn RN, Searle G, Abi-Dargham A, Slifstein M, Watson J, Laruelle M, Rabiner EA. An evaluation of the brain distribution of [(11)C]GSK1034702, a muscarinic-1 (M 1) positive allosteric modulator in the living human brain using positron emission tomography. EJNMMI Res. 2014 Dec;4(1):66. doi: 10.1186/s13550-014-0066-y. Epub 2014 Dec 5. PMID 26116126
- See also: Results for study 110771 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/110771?search=study&study_ids=110771#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 110771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110771 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register